CLINICAL TRIAL: NCT00008749
Title: Role of Altered CD40-Ligand Gene Transcription in Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Arthritis Foundation (Other)
Other Study IDs: NCRR-M01RR00240-1736
Record Dates: First submitted 2001-01-16; First posted 2001-01-18 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control

SUMMARY:
Systemic lupus erythematosus is an often devastating autoimmune disease which affects 1 in 2,000 women in the United States. Recently, several research laboratories have reported that a protein, named CD40-ligand (CD154), is overexpressed by a subset of white blood cells, called lymphocytes, in patients with lupus. Expression of CD154 appears critical to the generation of antibodies that cause disease in lupus. Blocking CD154 interactions in the immune system has been shown to decrease disease activity in animal models of lupus. We propose to study the regulation of CD154 in patients with lupus in hopes of inhibiting its abnormal and deleterious expression.

ELIGIBILITY:
Inclusion:

A diagnosis of systemic lupus erythematosus

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States